CLINICAL TRIAL: NCT04115852
Title: Investigating the Neural Correlates of Interoceptive Nutritional Processing Using fMRI in Healthy Participants and Patients With Binge-Eating-Disorder
Brief Title: Interoceptive Nutritional Processing in Healthy Participants and Patients With Binge-Eating-Disorder
Acronym: BAG-C
Status: Completed | Type: Observational
Sponsor: University of Heidelberg Medical Center (Other)
Responsible Party: Principal Investigator, Joe Simon, Principal Investigator, University of Heidelberg Medical Center
Other Study IDs: S-545/2019
Record Dates: First submitted 2019-10-02; First posted 2019-10-04 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: Food Habits; Binge-Eating Disorder
Keywords: fmri; interoceptive food processing
MeSH Terms: conditions — Feeding Behavior; Binge-Eating Disorder | interventions — CYFIP2 protein, human

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- CON: Healthy Controls
  Interventions: Behavioral: fmri
- BED: Patients with Binge-Eating-Disorder
  Interventions: Behavioral: fmri

INTERVENTIONS:
Behavioral: fmri — functional magnetic resonance imaging

SUMMARY:
Binge-Eating-Disorder (BED) is a common eating disorder characterized by recurring episodes of uncontrollable eating. The underlying neural mechanisms are largely unknown. However, dysfunctional hormonal satiety signaling as well as dysfunctional neural processing of food cues are discussed as possible casual factors in the development and maintenance of this disorder. Additional research is needed to specify the exact contribution of these observations and how they interact with each other. Accordingly, the current study plans to investigate metabolic gut-brain signaling to better understand the underlying causes of abnormal eating behavior. To this end, 25 healthy normal weight control participants as well as 25 patients with BED will be recruited. The responsivity of the hypothalamus (i.e., the core region of homeostatic control) and its interaction with the mesocorticolimbic reward system will be assessed by applying a single-blind, randomized, crossover design of intravenous infusion of glucose or NaCl. This approach allows the study of gut-brain signaling to the hypothalamus and the reward system by controlling for sensory aspects of food intake (sight, smell, and taste). The interaction between the hypothalamus and the mesocorticolimbic reward system will be investigated using an effective connectivity analysis. FMRI with high spatial resolution and with an optimized protocol for the investigation of the hypothalamus and the mesocorticolimbic reward system will be employed. A better understanding of the underlying psychobiological mechanisms of BED is a fundamental requirement for the development of improved prevention and treatment strategies

ELIGIBILITY:
Inclusion criteria:

1. patients that meet the diagnostic criteria for BED
2. Over age of 18 years.
3. Right-handedness.
4. Normal or corrected-to-normal vision.
5. No other lifetime or current medical illness that could potentially affect appetite or body weight

Exclusion criteria (for all participants):

1. History of head injury or surgery
2. History of neurological disorder
3. Severe psychiatric comorbidity (psychosis, bipolar disorder, substance abuse)
4. Smoking
5. Borderline personality disorder
6. Current psychotropic medication
7. Inability to undergo fMRI scan (e.g. metallic implants, claustrophobia, pacemakers)
8. Pregnancy

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will enroll 25 patients with BED. Patients will be recruited from the investigator's in- and out-patient department or by public advertisement after giving their written informed consent. Additionally, a healthy control group of 25 participants will be recruited by public advertisement.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
the neural correlates of interoceptive nutritional processing | 2-3 weeks
  cross-sectional fMRI

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Heidelberg, Heidelberg, Germany

IPD SHARING:
Plan to Share IPD: Undecided